CLINICAL TRIAL: NCT04390945
Title: Camrelizumab Combined With Concurrent Radiotherapy and Chemotherapy for Treatment of Patients With Local Recurrence of Esophageal Cancer
Brief Title: Camrelizumab Combined With CRT for Treatment of Patients With Local Recurrence of Esophageal Cancer
Status: Unknown | Phase: Phase 2 | Type: Interventional
Last Known Status: Recruiting
Sponsor: The First Affiliated Hospital of Henan University of Science and Technology (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: FirstHenanUST-EC
Record Dates: First submitted 2020-05-13; First posted 2020-05-18 (Actual); Last update posted 2022-02-03 (Actual); Status verified 2022-01

CONDITIONS: Esophageal Cancer
MeSH Terms: conditions — Esophageal Neoplasms | interventions — camrelizumab; Capecitabine

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Camrelizumab Combined With Concurrent Radiotherapy and Chemotherapy (Experimental): Camrelizumab (200mg Q2W, continuous medication until disease progression, intolerable toxicity, or withdrawal due to other reasons) Simultaneous radiotherapy (50-50.4Gy / 1.8-2Gy / 25-28F) Chemotherapy (Capecitabine, 625mg/m2, bid, oral, d1-5, qw, total 5 weeks).
  Interventions: Drug: Camrelizumab

INTERVENTIONS:
Drug: Camrelizumab — Camrelizumab combined with concurrent radiotherapy and chemotherapy
  Other Names: Capecitabine; concurrent radiotherapy

SUMMARY:
China is a country with a large incidence of esophageal cancer. The prevalence and mortality rate of esophageal cancer in China ranks fifth in the world. However, due to China's huge population base, new patients with esophageal cancer and deaths account for about 55% of the world. This study aimed to explore the efficacy and safety of Camrelizumab Combined With Concurrent Radiotherapy and Chemotherapy for Treatment of Patients With Local Recurrence of Esophageal Cancer.

DETAILED DESCRIPTION:
This is an open clinical study to evaluate the efficacy and safety of Camrelizumab combined with Concurrent Radiotherapy and Chemotherapy in the treatment of locally recurrent esophageal cancer.

Objective to study patients with local recurrence of esophageal cancer after radical treatment.

The study will take progression free survival (PFS) as the main efficacy index, and plan to enroll about 62 patients with local recurrence of esophageal cancer after radical treatment. After fully informed and signed the informed consent, the subjects will enter the experimental stage after screening.

ELIGIBILITY:
Inclusion Criteria:

1. Age 18-75 years old, both men and women;
2. Histologically confirmed as esophageal cancer;
3. Patients with local recurrence of esophageal cancer after radical treatment;
4. ECOG: 0 ～ 1;
5. Expected survival time ≥ 12 weeks;
6. The function of main organs is normal, that is, it meets the following standards:

(1) Blood routine examination:

a. HB≥90g / L; b.ANC≥1.5 × 109 / L; c.PLT≥80 × 109 / L; (2) Biochemical inspection:

a. ALB ≥ 30g / L; b. ALT and AST ≤ 2.5ULN; if there is liver metastasis, ALT and AST ≤ 5ULN; c. TBIL ≤ 1.5ULN; 7. Women of childbearing age should agree to use contraceptive measures (such as intrauterine devices, contraceptives or condoms) during the study period and within 6 months after the end of the study; the serum or urine pregnancy test is negative within 7 days before the study enrollment , and must be a non-lactating patient; males should agree to patients who must use contraception during the study period and within 6 months after the end of the study period; 8. Subjects voluntarily joined the study, signed an informed consent form, had good compliance, and cooperated with follow-up.

Exclusion Criteria:

1. Does not meet the above selection criteria;
2. Patients with distant visceral metastasis;
3. Patients with recurrence time <10 months receiving radical radiotherapy
4. Those who are allergic to or metabolic disorders of capecitabine and Camrelizumab;
5. The patient has any active autoimmune disease or has a history of autoimmune disease (such as the following, but not limited to: autoimmune hepatitis, interstitial pneumonia, uveitis, enteritis, hepatitis, pituitary inflammation, vasculitis, nephritis , Hyperthyroidism; The patient has vitiligo; Asthma has been completely relieved in childhood and can be included without any intervention after adulthood; Patients with asthma requiring medical intervention with bronchodilators cannot be included);
6. The patient is using immunosuppressive agents or systemic hormone therapy to achieve the purpose of immunosuppression (dose> 10mg / day prednisone or other therapeutic hormones), and is still using it within 2 weeks before enrollment
7. Contraindications to radiotherapy;
8. Severe infections that are active or uncontrolled;
9. Liver diseases such as decompensated liver disease, active hepatitis B (HBV-DNA≥104 copies / ml or 2000IU / ml) or hepatitis C (hepatitis C antibody is positive, and HCV-RNA is higher than the analytical method.
10. Patients whose imaging has shown that the tumor has invaded the important blood vessels or the investigator judges that the tumor is likely to invade the important blood vessels and cause fatal hemorrhage during the follow-up study;
11. Pregnant or lactating women;
12. Patients with other malignant tumors within 5 years (except basal cell carcinoma of the skin and cervical carcinoma in situ);
13. Patients with a history of psychotropic substance abuse who are unable to quit or have mental disorders;
14. Patients who have participated in clinical trials of other drugs within four weeks;
15. According to the judgment of the investigator, there are patients with concomitant diseases that seriously endanger the safety of the patient or affect the completion of the study;
16. The investigator considers it unsuitable for inclusion.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 62 (Estimated)
Dates: Start 2021-12-01 (Actual); Primary Completion 2023-10 (Estimated); Study Completion 2024-08 (Estimated)

PRIMARY OUTCOMES:
Progression-free survival，PFS | 9 months
  Time from randomization to patient's tumor progression or death

SECONDARY OUTCOMES:
Overall survival，OS | 1 year
  The time from the beginning of randomization to death due to any cause.
Objective Response Rate, ORR | 1 year
  The proportion of patients whose tumor shrinks to a certain amount and remains for a certain period of time

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Henan University of Science and Technology, Luoyang, Henan, China